CLINICAL TRIAL: NCT06465849
Title: Clinical Evaluation of the Effect of Reduced Dentin Etching Time Using Two Universal Adhesives in Restorations of Non-carious Cervical Lesions: Double-blind Randomized Clinical Trial
Brief Title: Evaluation of the Reduced Dentin Etching Time Using Universal Adhesives in the Quality of Cervical Lesions Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Agencia Nacional de Investigación y Desarrollo (Other)
Responsible Party: Principal Investigator, Mario Felipe Gutiérrez Reyes, Associate Professor, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEC2024055
Record Dates: First submitted 2024-06-13; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Non-carious Cervical Lesions
Keywords: Dental bonding; Tooth erosion; Tooth Wear; Adhesive systems; Etching Time
MeSH Terms: conditions — Tooth Erosion; Tooth Wear

STUDY DESIGN:
Intervention Model Description: This is a four-arm, double-blind, randomized controlled clinical trial. Experimental group 1: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (3M) on dentin etched for 5 seconds.
  Experimental group 2: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Kulzer) on dentin etched for 5 seconds.
  Control group 1: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (3M) on dentin etched for 15 seconds.
  Control group 2: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Kulzer) on dentin etched for 15 seconds.
  LCNCs will be randomized to universal adhesive usage and etching time.
Who Masked: Participant, Outcomes Assessor
Masking Description: Two blinded, experienced, and calibrated dentists (who specialized in esthetic dentistry with more than 15 years of clinical practice), will perform the clinical evaluation. Patients will be also blinded to group assignment. An inter-examiner and inter-examiner agreement of at least 85% will be necessary before beginning the evaluation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1 (Experimental): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations in the etch-and-rinse strategy.
  Interventions: Procedure: Dentin Etching time for 5 seconds; Device: Scotchbond Universal Plus; 3M
- Experimental group 2 (Experimental): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations in the etch-and-rinse strategy.
  Interventions: Procedure: Dentin Etching time for 5 seconds; Device: Gluma Universal Bond; Kulzer
- Control group 1 (Active Comparator): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations in the etch-and-rinse strategy.
  Interventions: Device: Scotchbond Universal Plus; 3M; Procedure: Dentin Etching time for 15 seconds
- Control group 2 (Active Comparator): 35 non-carious cervical lesions (NCCL) will receive composite resin restorations in the etch-and-rinse strategy.
  Interventions: Device: Gluma Universal Bond; Kulzer; Procedure: Dentin Etching time for 15 seconds

INTERVENTIONS:
Procedure: Dentin Etching time for 5 seconds — Composite resin restorations of non-carious cervical lesions will be performed with an adhesive on dentin etched for 5 seconds in the etch-and-rinse application strategy.
  Arms: Experimental group 1; Experimental group 2
Device: Scotchbond Universal Plus; 3M — Composite resin restorations of non-carious cervical lesions will be performed with an universal adhesive (Scotchbond Universal Plus; 3M).
  Arms: Control group 1; Experimental group 1
Device: Gluma Universal Bond; Kulzer — Composite resin restorations of non-carious cervical lesions will be performed with an universal adhesive (Gluma Universal Bond; Kulzer).
  Arms: Control group 2; Experimental group 2
Procedure: Dentin Etching time for 15 seconds — Composite resin restorations of non-carious cervical lesions will be performed with an adhesive on dentin etched for 15 seconds in the etch-and-rinse application strategy.
  Arms: Control group 1; Control group 2

SUMMARY:
The aim of this study will be to evaluate the effect of reduced dentin etching time on the 6- and 12-months clinical performance of two universal adhesive systems used as etch-and-rinse application mode in non-carious cervical lesions (NCCLs).

Materials & Methods: 140 restorations will be randomly placed in 35 subjects according to the following groups: SUP5 (Scotchbond Universal Plus adhesive on dentin etched for 5 seconds); SUP15 (Scotchbond Universal Plus adhesive on dentin etched for 15 seconds); GBU5 (Gluma Universal Bond adhesive on dentin etched for 5 seconds); GBU15 (Gluma Universal Bond adhesive on dentin etched for 15 seconds). All groups will be light-cured for 10s/1,000 mW/cm2. A resin composite will be placed by applying three increments and each one will be light cured for 20s/1,000 mW/cm2. The restorations will be finished immediately with fine diamond burs and polishers. The restorations will be evaluated at baseline and after 6- and 12-months by using the FDI criteria. The following outcomes will be evaluated: retention, marginal staining, marginal adaptation, post-operative sensitivity and recurrence of caries. The differences among the groups will be calculated using Friedman repeated measures analysis of variance rank (α = 0.05).

DETAILED DESCRIPTION:
This is a four-arm, double-blind, randomized controlled clinical trial. Experimental group 1: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Scotchbond Universal Plus; 3M) on dentin etched for 5 seconds in the etch-and-rinse application strategy.

Experimental group 2: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Gluma Universal Bond; Kulzer) on dentin etched for 5 seconds in the etch-and-rinse application strategy.

Control group 1: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Scotchbond Universal Plus; 3M) on dentin etched for 15 seconds in the etch-and-rinse application strategy.

Control group 2: 35 non-carious cervical lesions (NCCL) will receive composite resin restorations using an universal adhesive (Gluma Universal Bond; Kulzer) on dentin etched for 15 seconds in the etch-and-rinse application strategy.

LCNCs will be randomized to universal adhesive usage and dentin etching time. All groups will be light-cured with a lightcuring device (SmartLite Focus, Dentsply) with a light intensity of 900 mW/cm² for 10 seconds. Operators will restore the cervical area by applying three increments of resin (Vittra APS, FGM Prod. Odont.Ltda, Joinville, SC, Brazil). Each increment will light cure for 20 s at 900 mW/cm2 (SmartLite Focus, Dentsply). Restorations will be finished immediately with fine and extra fine diamond burs and polished with polishing gums.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Presence of at least two Non-Carious Cervical Lesions in the dental arch with a need for restorative treatment.
* Acceptable level of oral hygiene according to the Simplified Oral Hygiene Index.
* At least 20 teeth in function.
* Non-Carious Cervical Lesions with a maximum of 50% of enamel margin.

Exclusion Criteria:

* Driving difficulties that prevent adequate oral hygiene.
* Periodontal disease.
* Active caries lesions on the teeth included in the research.
* Parafunctional habits.
* Active staples of removable partial dentures on the teeth included in the research and that these are not pillars of prostheses.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Retention of restorations | From date of randomization until twenty four months
  Retention measured by World Dental Federation (FDI) criteria as following:
  * VG: Clinically very good - Restoration retained, no fractures / cracks;
  * G: Clinically good - Small hairline crack;
  * SS: Clinically sufficient/satisfactory - Two or more or larger hairline cracks and/or chipping (not affecting the marginal integrity);
  * US: Clinically unsatisfactory - Chipping fractures which damage marginal quality; bulk fractures with or without partial loss (less than half of the restoration);
  * PO: Clinically poor - (Partial or complete) loss of restoration, (replacement necessary).

SECONDARY OUTCOMES:
Marginal Adaptation of restorations | From date of randomization until twenty four months
  Marginal Adaptation measured by World Dental Federation (FDI) criteria as following:
  * VG: Clinically very good - Harmonious outline, no gaps, no discoloration;
  * G: Clinically good - Small marginal fracture removable by polishing;
  * SS: Clinically sufficient/satisfactory - Several small enamel or dentin fractures;
  * US: Clinically unsatisfactory - Notable enamel or dentine wall fracture;
  * PO: Clinically poor - Filling is loose but in situ.
Marginal Staining of restorations | From date of randomization until twenty four months
  Marginal Staining measured by World Dental Federation (FDI) criteria as following:
  * VG: Clinically very good - No marginal staining;
  * G: Clinically good - Minor marginal staining, easily removable by polishing;
  * SS: Clinically sufficient/satisfactory - Moderate marginal staining, not esthetically unacceptable;
  * US: Clinically unsatisfactory - Pronounced marginal staining; major intervention necessary for improvement;
  * PO: Clinically poor - Deep marginal staining not accessible for intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mario Felipe Gutiérrez Reyes, PhD, Study Director — Universidad de los Andes, Chile
Locations (1):
- Mario Felipe Gutiérrez Reyes, Santiago, Santiago Metropolitan, Chile